CLINICAL TRIAL: NCT05102877
Title: The Effect of Sensory Level Versus Motor Level Electrical Stimulation of Pharyngeal Muscles in Acute Stroke Patients With Dysphagia
Brief Title: Sensory Versus Motor Level Neuromuscular Electrical Stimulation
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Responsible Party: Principal Investigator, Emily Rosario, Director of Research, Casa Colina Hospital and Centers for Healthcare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMES 1.1
Record Dates: First submitted 2021-10-12; First posted 2021-11-02 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Stroke, Ischemic
Keywords: Dysphagia; Swallow; Stimulation
MeSH Terms: conditions — Ischemic Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sensory level stimulation (Experimental): ten, 45-minute anterior neck sensory level electrical stimulation sessions in addition to traditional dysphagia therapy.
  Interventions: Device: Neuromuscular electrical stimulation
- Motor level stimulation (Experimental): ten, 45-minute anterior neck sensory level electrical stimulation sessions in addition to traditional dysphagia therapy.
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Motor stimulation was administered at an intensity sufficient to produce muscle contractions. Sensory stimulation was defined as the threshold when the patient feels a tingling sensation on their skin.

SUMMARY:
Dysphagia is a serious cause of morbidity and mortality in stroke survivors. Electrical stimulation is often included as part of the treatment plan for dysphagia, and can be applied at a sensory or motor level intensity. However, evidence to support these different modes of stimulation is lacking. This study compared the effectiveness of sensory and motor level stimulation on post-stroke dysphagia.

DETAILED DESCRIPTION:
Objective: Dysphagia is a serious cause of morbidity and mortality in stroke survivors. Electrical stimulation is often included as part of the treatment plan for dysphagia, and can be applied at a sensory or motor level intensity. However, evidence to support sensory versus motor stimulation is lacking. This study compares the effect of sensory and motor stimulation on post-stroke dysphagia.

Design: Randomized controlled trial

Setting: Inpatient rehabilitation facility.

Participants: Participants (50-75 years of age) who had dysphagia caused by a stroke within 6 months prior to enrollment were included. Participants were excluded if they had a contraindication for electrical stimulation, previous stroke, psychiatric disorder, contraindications for MBS, or pre-stroke swallowing disorders.

Interventions: Each patient received ten, 45-minute anterior neck sensory or motor level electrical stimulation sessions in addition to standard speech therapy. Motor stimulation was administered as a stimulus intensity sufficient to produce muscle contractions. Sensory stimulation was defined as the threshold when the patient feels a tingling sensation on their skin (approximately 4-5mA).

Main Outcome Measures: Swallow FIM, National Outcome Measurement System (NOMS), Dysphagia Outcome Severity Scale (DOSS), and change in modified diet.

ELIGIBILITY:
Inclusion Criteria:

* 18-80
* acute ischemic CVA within the first month and confirmed by MRI.
* Diagnosis of dysphagia will be obtained by bedside swallowing exam and MBS/FEES studies.

Exclusion Criteria:

* patients who have contraindications for electrical stimulation (malignancy, DVT/thrombophlebitis, hemorrhagic conditions, pregnancy, pacemaker or other electrical hardware)
* known premorbid swallowing disorders
* GERD
* dementia or psychiatric disorder
* bilateral cerebral involvement
* contraindications for FEES/MBS (infectious disease such as HIV, HCV, HBV, nasal obstruction, decompensated heart disease, risk of bleeding such as active ulcers, allergy to contrast).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Swallow Functional Assessment Measure | up to 2 months
  7 point swallow scale the Functional oral intake scale (FOIS) lowest score = 1; highest = 7.
Change in Dysphagia outcome Severity Scale | up to 2 months
  seven-point functional outcome scale designed to assess dysphagia severity on the MBSS, lowest score = 1; highest = 7.

SECONDARY OUTCOMES:
Change in PenAsp | up to 2 months
  Evaluates the depth response and clearance of material entering into the airway, lowest score = 8; highest =1.
Change in Swal-Qol | up to 3 months
  93-item outcome tool 24 was used to determine impact on quality-of-life and quality-of-care. Each item has a 5 point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Emily R. Rosario, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare
Locations (1):
- Casa Colina Hospital and Centers for Healthcare, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No